CLINICAL TRIAL: NCT01217099
Title: A Prospective, Open-label Trial of Methylprednisolone Pulse Macrolide Therapy for Refractory Mycoplasma Pneumoniae Pneumonia in Children
Brief Title: Methylprednisolone Pulse Macrolide Therapy for Refractory Mycoplasma Pneumoniae Pneumonia in Children
Acronym: MPP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated
Sponsor: Chongqing Medical University (Other)
Responsible Party: zhengxiu luo, Children's Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR-TRC2
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2007-05

CONDITIONS: Refractory Mycoplasma Pneumoniae Pneumonia
Keywords: refractory mycoplasma pneumoniae pneumonia
MeSH Terms: conditions — Pneumonia, Mycoplasma | interventions — Methylprednisolone; Azithromycin; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylprednisolone (No Intervention): methylprednisolone pulse azithromycin
  Interventions: Drug: methylprednisolone
- azithromycin (No Intervention): azithromycin
  Interventions: Drug: azithromycin

INTERVENTIONS:
Drug: methylprednisolone — treatment patients were iv methylprednisolone pulse azithromycin for 5 days.
  Other Names: treatment group
  Arms: methylprednisolone
Drug: azithromycin — control patients were iv azithromycin for 5 days.
  Other Names: control group
  Arms: azithromycin

SUMMARY:
The purpose of this study is planned to investigate whether small doses of methylprednisolone pulse macrolide therapy can relieve symptoms,chest X-rays faster than macrolide alone therapy for refractory mycoplasma pneumoniae pneumonia(MPP) .

DETAILED DESCRIPTION:
Corticosteroid has been used in adulthood refractory MPP with satisfactory efficacy. But there were few studies about the use of corticosteroid in children with refractory MPP. Lee KY et al indicated oral prednisolone of 1 mg/kg/ day for 1 week be useful for children with severe MPP. Akihiro T et al demonstrated that intravenously administered methylprednisolone at a dose of 30 mg/kg once daily for 3 consecutive days had an efficacious treatment for children with refractory MPP.But the methods of corticosteroid use, such as the dosage, administration route, duration of treatment have not been well understood. So in this study, we planned to investigate whether small doses of methylprednisolone pulse macrolide therapy can relieve symptoms,chest X-rays faster than macrolide alone therapy for refractory mycoplasma pneumoniae pneumonia in a prospective, open-label fashion.

PMID: 11096025 PMID: 18033831 PMID: 10434547 PMID: 16437541 PMID: 18656264

ELIGIBILITY:
Inclusion Criteria:

* mycoplasma pneumoniae pneumonia
* prolonged fever and deterioration of radiological findings despite macrolides treatment for 7 days or more.

Exclusion Criteria:

* chronic cardiac and pulmonary disease
* immunodeficiency
* requiring mechanical ventilation
* with other pathogens detected during pneumonia.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2007-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
efficacy of methylprednisolone pulse macrolide therapy for children with refractory MPP. | 3-year
  compare the temperature , infiltration absorption,atelectasis resolution, pleural effusion disappearance,serum levels of ferritin and LDH between methylprednisolone pulse macrolide therapy group and macrolide therapy group .

SECONDARY OUTCOMES:
safety of methylprednisolone pulse macrolide therapy for children with refractory MPP. | 3-year
  observe the further complications of infection between methylprednisolone pulse macrolide therapy group and macrolide therapy group .

CONTACTS AND LOCATIONS:
Overall Officials: zhengxiu luo, doctor, Principal Investigator — Chongqing Medical University

REFERENCES:
- See also: Related Info — http://www.clinicaltrials.gov